CLINICAL TRIAL: NCT02543528
Title: Echo Ionic Silicone Hydrogel 6-Month Extended Wear Investigation
Brief Title: A Clinical Trial to Evaluate Investigational Silicone Hydrogel Contact Lenses Worn Continuously for One Week
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5201
Record Dates: First submitted 2015-08-06; First posted 2015-09-07 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Visual Disorder
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- etafilcon A (1-Day) and etafilcon A (Reusable) (Experimental): Prior to randomization, all subjects will participate in a 2-week contact lens adaptation period wearing etafilcon A (1-Day). Subjects will then be randomized to one of four experimental contact lenses to be worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Interventions: Device: etafilcon A (Reusable); Device: etafilcon A (1-Day)
- etafilcon A (1-Day) and Investigational Lens 1 (Experimental): Prior to randomization, all subjects will participate in a 2-week contact lens adaptation period wearing etafilcon A (1-Day). Subjects will then be randomized to one of four experimental contact lenses to be worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Interventions: Device: Investigational Lens 1; Device: etafilcon A (1-Day)
- etafilcon A (1-Day) and Investigational Lens 2 (Experimental): Prior to randomization, all subjects will participate in a 2-week contact lens adaptation period wearing etafilcon A (1-Day). Subjects will then be randomized to one of four experimental contact lenses to be worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Interventions: Device: Investigational Lens 2; Device: etafilcon A (1-Day)
- etafilcon A (1-Day) and Investigational Lens 3 (Experimental): Prior to randomization, all subjects will participate in a 2-week contact lens adaptation period wearing etafilcon A (1-Day). Subjects will then be randomized to one of four experimental contact lenses to be worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Interventions: Device: Investigational Lens 3; Device: etafilcon A (1-Day)

INTERVENTIONS:
Device: Investigational Lens 1 — One fresh pair of Investigational Lens 1 contact lenses worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Arms: etafilcon A (1-Day) and Investigational Lens 1
Device: Investigational Lens 2 — One fresh pair of Investigational Lens 2 contact lenses worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Arms: etafilcon A (1-Day) and Investigational Lens 2
Device: Investigational Lens 3 — One fresh pair of Investigational Lens 3 contact lenses worn continuously in 6 nights/7 days wear cycles for 6 months of total wear.
  Arms: etafilcon A (1-Day) and Investigational Lens 3
Device: etafilcon A (Reusable) — One fresh pair of etafilcon A (Reusable) contact lenses worn continuously in 6nights/7 days wear cycles for 6 months of total wear.
  Arms: etafilcon A (1-Day) and etafilcon A (Reusable)
Device: etafilcon A (1-Day) — 2-week contact lens adaptation period wearing prior to randomization

SUMMARY:
This study is a prospective, randomized, double-masked, bilateral, dispensing, parallel-group clinical trial design. All subjects will participate in a 2-week daily disposable contact lens adaptation period prior to being randomized into one of the four extended wear lenses. The study has a total of 9 scheduled study visits and a total duration of ~197 days. The lenses will be replaced with a fresh pair after 6 nights / 7 days of wear.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read and understand English and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 and no more than 39 years of age.
* The subject's spherical equivalent distance refraction must be in the range of -1.00 to -5.50 diopters in each eye.
* The subject's refractive cylinder must be less than 1.00 diopters in each eye.
* The subject must have best corrected visual acuity of 20/30 or better in each eye.
* The subject must be without history of contact lens use in the past 12 months.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

* Any previous experience wearing contact lenses on an overnight or extended wear basis (at least 1 night per month)
* Currently pregnant or lactating (self reported) (subjects who become pregnant during the study will be discontinued).
* Currently a regular smoker (1 or more times per month).
* Current routine swimmer (1 or more times per month).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease (ex. Sjögren's Syndrome), autoimmune disease (ex. rheumatoid arthritis), or use of medication (ex. chronic steroid use), which may interfere with contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
* Any previous or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser in situ keratomileusis (LASIK), etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV) by self report).
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Foundation, Sankara Nethralaya, Chennai, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study utilized an adaptation period of 14 days prior to dispensing the extended wear contact lenses. A total of 171 subjects were enrolled into the adaption period. Of those enrolled into this period 168 were dispensed a study lens and 3 did not meet the eligibility criteria. Of the 168 dispensed subjects 142 completed the adaptation period.
Pre-assignment Details: A total of 26 subjects were discontinued from the adaptation period. A total of 142 subjects were enrolled into the extended wear period. Of the enrolled subjects, all 142 were dispensed a study lens. Of the dispensed subjects in the extended wear period 58 completed the study and 84 subjects discontinued from the study.
Groups:
- Investigational Lens 1: Subjects that were randomized to receive the investigational contact lens 1 throughout the entire duration of the extended wear period.
- Investigational Lens 2: Subjects that were randomized to receive the investigational contact lens 2 throughout the entire duration of the extended wear period.
- Investigational Lens 3: Subjects that were randomized to receive the investigational contact lens 3 throughout the entire duration of the extended wear period.
- Etafilcon A (Resuable): Subjects that were randomized to receive the etafilcon A (Reusable) lens throughout the entire duration of the extended wear period.
- Etafilcon A (1-Day): All subjects wore the etafilcon A 1-Day contact lens during the 2-week adaptation period.
Period: Adaptation Period
Arm/Group | Investigational Lens 1 | Investigational Lens 2 | Investigational Lens 3 | Etafilcon A (Resuable) | Etafilcon A (1-Day)
Started (168) | 0 | 0 | 0 | 0 | 168
Completed (142) | 0 | 0 | 0 | 0 | 142
Not Completed | 0 | 0 | 0 | 0 | 26
Not completed — Unsatisfactory Lens Fitting | 0 | 0 | 0 | 0 | 2
Not completed — Lens Handling Difficultes | 0 | 0 | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Period: Extended Wear Period
Arm/Group | Investigational Lens 1 | Investigational Lens 2 | Investigational Lens 3 | Etafilcon A (Resuable) | Etafilcon A (1-Day)
Started | 36 | 35 | 36 | 35 | 0
Completed | 8 | 14 | 13 | 23 | 0
Not Completed | 28 | 21 | 23 | 12 | 0
Not completed — Adverse Event | 17 | 11 | 16 | 3 | 0
Not completed — Missed too many scheduled visits | 0 | 0 | 1 | 3 | 0
Not completed — Unsatisfactory Lens Fitting | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 10 | 9 | 4 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed at least 1 study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All subjects enrolled into the adaptation or extended wear period of the study.
  Years | 20.2 (2.80)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: All subjects enrolled into the adaptation or extended wear period of the study.
  Participants
    Female | 108
    Male | 60
Race/Ethnicity, Customized [Number; unit: Participants] — Population: All subjects that were enrolled into the adaptation or extended wear period of the study.
  Participants
    Asian Indian | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of First Occurred Serious and Significant Lens-related Corneal Infiltrative Event (CIE)
Description: The number of first serious and significant corneal infiltrative adverse events deemed to be related to contact lens wear (possible, probable or very likely) during a 6-month period (contact lens extended wear period) was assessed via Biomicroscopy. A biomicroscope was used to detect the presence of a corneal infiltrate for each subject eye (Yes: corneal infiltrates detected, No: None present). The number of subjects with corneal infiltrative events was reported for each lens type.
Time Frame: Up to 6 months
Population: The analysis population consists of all subjects that were enrolled into the extended wear period.
Measure: Number; unit: Number of Events
Units Other Than Participants: Eyes
Groups:
- Etafilcon A (Resuable): Subjects that were randomized to received the etafilcon A (Reusable) lens throughout the entire duration of the extended wear period.
Arm/Group | Investigational Lens 1 | Investigational Lens 3 | Investigational Lens 2 | Etafilcon A (Resuable)
Number analyzed (Participants) | 36 | 36 | 35 | 35
Number analyzed (Eyes) | 72 | 72 | 70 | 70
Number of Events | 14 | 13 | 12 | 1

2. Secondary Outcome: Overall Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience (CLUE)TM questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD). CLUE was collected at the 1-day, 5-day, 12-day, 26-day, 88-day and 180-day follow-up evaluation.
Time Frame: Time Frame Up to 6 months
Population: The analysis population consists of all subjects that have completed all study visits without a major protocol deviation in both the adaptation and extended wear periods.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Investigational Lens 3; Investigational Lens 1: Subjects that were randomized to receive the investigational contact lens 1 throughout the entire duration of the extended wear period.
Arm/Group | Investigational Lens 3 | Investigational Lens 1 | Investigational Lens 2 | Etafilcon A (Resuable)
Number analyzed (Participants) | 8 | 13 | 14 | 23
Units on a Scale
  1-Day Follow-up | 59.39 (14.263) | 60.22 (9.005) | 58.85 (13.102) | 62.51 (13.431)
  5-Day Follow-up | 58.38 (9.293) | 60.12 (8.447) | 58.29 (9.735) | 64.59 (13.301)
  12-Day Follow-up | 60.94 (9.620) | 65.74 (12.091) | 58.95 (13.457) | 64.87 (13.831)
  26-Day Follow-up | 60.20 (12.851) | 65.41 (16.467) | 57.35 (15.280) | 65.57 (14.513)
  88-Day Follow-up | 59.54 (7.474) | 55.59 (15.247) | 57.71 (12.150) | 65.00 (15.657)
  180-Day Follow-up | 57.81 (9.133) | 62.69 (14.600) | 54.91 (7.578) | 64.49 (16.120)

3. Secondary Outcome: Overall Vision Score
Description: Overall quality of vision score was assessed using the Contact Lens User Experience (CLUE)TM questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD). CLUE was collected at the 1-day, 5-day, 12-day, 26-day, 88-day and 180-day follow-up evaluation.
Time Frame: Time Frame Up to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Investigational Lens 3 | Investigational Lens 1 | Investigational Lens 2 | Etafilcon A (Resuable)
Number analyzed (Participants) | 8 | 13 | 14 | 23
Units on a Scale
  1-Day Follow-up | 55.27 (15.819) | 56.78 (14.299) | 52.87 (12.857) | 60.28 (14.723)
  5-Day Follow-up | 53.02 (9.117) | 54.66 (14.398) | 52.11 (13.284) | 59.55 (15.169)
  12-Day Follow-up | 52.17 (13.614) | 59.63 (17.147) | 50.73 (11.715) | 59.59 (14.892)
  26-Day Follow-up | 52.85 (5.218) | 57.84 (13.257) | 50.38 (17.434) | 59.76 (14.244)
  88-Day Follow-up | 50.23 (17.080) | 54.22 (14.718) | 50.67 (10.777) | 63.83 (17.096)
  180-Day Follow-up | 53.49 (9.883) | 54.07 (10.654) | 50.92 (9.699) | 61.68 (16.426)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 6 months per subject.
Groups:
- Etafilcon A (1-Day): All subject wore the etafilcon A (1-Day) contact lens throughout the entire duration of the adaptation period (14-Days).
Arm/Group | Etafilcon A (1-Day) | Investigational Lens 1 | Investigational Lens 2 | Investigational Lens 3 | Etafilcon A (Resuable)
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/36 | 0/35 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/36 | 0/35 | 3/36 | 1/35
Other Adverse Events (participants affected / at risk) | 12/168 | 36/36 | 27/35 | 33/36 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etafilcon A (1-Day) (N=168) | Investigational Lens 1 (N=36) | Investigational Lens 2 (N=35) | Investigational Lens 3 (N=36) | Etafilcon A (Resuable) (N=35)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etafilcon A (1-Day) (N=168) | Investigational Lens 1 (N=36) | Investigational Lens 2 (N=35) | Investigational Lens 3 (N=36) | Etafilcon A (Resuable) (N=35)
Fever (Immune system disorders) | 5 (5) | 2 (2) | 4 (4) | 1 (1) | 6 (6)
CLPC (Contact Lens Papillary Conjunctivitis) (Eye disorders) | 0 (0) | 2 (4) | 2 (3) | 2 (3) | 0 (0)
Meibomianitis (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
NSIE (Non-significant Infiltrative Event) (Eye disorders) | 1 (2) | 2 (2) | 5 (5) | 4 (4) | 2 (2)
Corneal Foreign Body (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Slit Lamp Findings Grade 2 or less requiring treatment (Eye disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 2 (2)
SPK (Superficial Punctate Keratitis) (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Symptoms Problems or Complaints Requiring Treatment (Eye disorders) | 1 (1) | 6 (6) | 3 (3) | 3 (3) | 4 (7)
CLPU (Contact Lens induced Peripheral Ulcer) (Eye disorders) | 0 (0) | 12 (12) | 10 (10) | 10 (12) | 0 (0)
Asymptomatic Corneal Scar (Eye disorders) | 0 (0) | 6 (8) | 7 (9) | 6 (8) | 5 (5)
SIE (Significant Infiltrative Event) (Eye disorders) | 0 (0) | 1 (2) | 4 (5) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days